CLINICAL TRIAL: NCT05988268
Title: Comparison of the Effects of 6-Week Vibration and Non-Vibration Foam Rolling on Neuromuscular Control and Performance in Male Soccer Players
Brief Title: Effects of 6-Week Vibration and Non-Vibration Foam Rolling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Celal Bayar University (Other)
Collaborators: Izmir Katip Celebi University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CBU-FTR-ES-O3
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Healthy Volunteers
Keywords: Physical fitness; Athletic Performance; Sports; Rehabilitation

STUDY DESIGN:
Intervention Model Description: Three groups as follows: Vibration Foam Rolling Group, Non-Vibration Foam Rolling Group, and Control Group
Who Masked: Participant, Outcomes Assessor
Masking Description: The control group will receive a routine warm-up protocol. Outcome measurement will be performed by an investigator who was blinded to group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Vibration Foam Rolling Group (Active Comparator): The vibration foam rolling method will be applied to the gluteal, tensor fascia latae, hamstring, quadriceps femoris, and gastrocnemius muscles of both lower extremities of the participants in the Vibration Foam Rolling Group, in addition to the routine warm-up protocol, 3 days a week for a total of 15 minutes a day for 6 weeks.
  Interventions: Other: Vibration Foam Rolling
- Non-Vibration Foam Rolling Group (Active Comparator): The non-vibration foam rolling method will be applied to the gluteal, tensor fascia latae, hamstring, quadriceps femoris, and gastrocnemius muscles of both lower extremities of the participants in the Non-Vibration Foam Rolling Group, in addition to the routine warm-up protocol, 3 days a week for a total of 15 minutes a day for 6 weeks.
  Interventions: Other: Non-Vibration Foam Rolling
- Control Group (No Intervention): No intervention will be applied to the control group. This group will continue the routine warm-up protocol.

INTERVENTIONS:
Other: Vibration Foam Rolling — The vibration foam rolling method will be applied to the gluteal, tensor fascia latae, hamstring, quadriceps femoris, and gastrocnemius muscles of both lower extremities of the participants in the Vibration Foam Rolling Group, in addition to the routine warm-up protocol, 3 days a week for a total of 15 minutes a day for 6 weeks.
  Arms: Vibration Foam Rolling Group
Other: Non-Vibration Foam Rolling — The non-vibration foam rolling method will be applied to the gluteal, tensor fascia latae, hamstring, quadriceps femoris, and gastrocnemius muscles of both lower extremities of the participants in the Non-Vibration Foam Rolling Group, in addition to the routine warm-up protocol, 3 days a week for a total of 15 minutes a day for 6 weeks.
  Arms: Non-Vibration Foam Rolling Group

SUMMARY:
This study aims to compare the effects of 6-week vibration and non-vibration foam rolling on neuromuscular control and performance in male soccer players.

DETAILED DESCRIPTION:
The typical warm-up protocol consists of different stretching exercises, sub-maximal aerobic activities, and sports-related activities. However, in recent years, warm-up protocols involving different methods have been applied and recommended.

Foam rolling (FR) via foam roller, one of these methods, has become a common and popular method in many sports settings.

While the popularity and use of the foam rolling method is gradually increasing, in recent years this method has begun to be applied as vibration and included in warming protocols.

The aim of this study is to compare the effects of 6-week vibration and non-vibration foam rolling on neuromuscular control and performance in male soccer players.

Within the scope of initial assessments; knee flexor and extensor muscle strength and Hamstring/Quadriceps muscle strength ratio with the Lafayette manual muscle testing device, flexibility with the sit-and-reach test, dynamic balance with the Y balance test, reaction time with the "Test You Brain Pro System", lower extremity anaerobic power with the Wingate anaerobic power test, agility with the t-test and sprint with the 20-m sprint test will be evaluated.

After the initial assessment, vibration and non-vibration foam rolling methods will be applied to the gluteal, tensor fascia latae, hamstring, quadriceps femoris and gastrocnemius muscles of both lower extremities of the participants in the intervention groups, in addition to the routine warm-up protocol, 3 days a week for a total of 15 minutes a day for 6 weeks. No intervention will be applied to the participants in the control group. This group will continue the routine warm-up protocol.

After the methods applied to the intervention groups for 6 weeks, the initial assessments applied to all participants will be repeated.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study.
* To regularly participate in team training within the club.
* To have been playing football for at least 1 year in the category.

Exclusion Criteria:

* Having any sports injury involving the lower extremity and/or spine in the last 3 months.
* Having a problem (vertigo, neuropathy, etc.) that may negatively affect balance and coordination.
* Having a musculoskeletal deformity (short limb, etc.) concerning the lower and upper extremities.
* Implementing a training program outside of routine team training

Ages: 18 Years to 22 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2023-08-07 (Actual); Primary Completion 2023-09-25 (Actual); Study Completion 2023-10-02 (Actual)

PRIMARY OUTCOMES:
Knee Flexor and Extensor Muscle Strength | A week
  Participants' knee flexor and extensor muscle strength will be evaluated with the Lafayette manual muscle test device (Lafayette Instrument Company, Lafayette IN, USA).This device is a valid and reliable method that is frequently used in the evaluation of muscle strength.
  During the evaluation, participants will be asked to perform a maximum isometric contraction for 3 seconds with the muscle in which the muscle strength is evaluated against the resistance to be applied with the manual muscle test device. Measurements will be repeated 3 times with one minute intervals for the right and left sides and the average of the measured values will be used for analysis.
Knee Flexor and Extensor Muscle Strength Ratio (H/Q Ratio) | A week
  Participants' Hamstring/Quadriceps muscle strength ratio will be evaluated with the Lafayette manual muscle test device (Lafayette Instrument Company, Lafayette IN, USA). This device is a valid and reliable method that is frequently used in the evaluation of muscle strength. The Hamstring/Quadriceps muscle strength ratio will be determined by the ratio of the knee flexor and extensor muscle strengths obtained during the measurements.
Flexibility | A week
  The flexibility will be evaluated whit the sit-and-reach test. The testing box will be fixed to the wall, and participants will be requested to sit with their knees extended and the soles of their feet against the testing box. Then participants will be requested to slowly reach forward as far as possible along the top of the box and hold the position for 2 seconds without bending their knees. The average of the two trials will be used for analysis.

SECONDARY OUTCOMES:
Dynamic Balance | A week
  Dynamic balance will be evaluated with the Y balance test. The test is a valid and reliable method that was developed as a version of the Star Excursion Balance Test (SEBT) to improve repeatability and standardize the performance. During the preparation of the test, three tape measures; between the anterior and the posterolateral/posteromedial directions, will be fixed to the ground with 135° angles. The measurement will be done for the dominant side three times after the trial and the average of the endpoints where the athletes could reach will be used for analysis. The greater the distance the participants can reach during the test, the better participant's dynamic balance performance.
Agility | A week
  Agility will be evaluated with the agility T-test. The test is a valid and reliable method used in the assessment of agility performance. For this test, an agility circuit will be created with 4 cones named 1, 2, 3, and 4. Cones will also set up at a distance of 10 yards between 1 and 2, and 5 yards between 2, and 3, 2, and 4. At the "go" command, the participant will sprint forward from cone 1 to cone 2, sidestepped to cone 3, sidestepped to cone 4, sidestepped to cone 2, then backpedal as fast as possible to cone 1. A stopwatch will be used during the test. The test will be performed 2 times with at least 2-minute rest periods between trials. The average of the 2 trials will be used for data analysis.
Sprint | A week
  Sprint performance will be evaluated with the 20-m sprint test. The test is a valid and reliable method used in studies to evaluate sprint performance. During the test, at the "go" command, the participant will be asked to complete the 20-meter distance as quickly as possible, and a stopwatch will be used to determine the time to complete the test. All participants will performed the test 2 times with at least 2-minute rest periods between trials. The average of the 2 trials will be used for data analysis.
Reaction Time | A week
  Lower-extremity V-MRT will be evaluated with the Test You Brain Pro System. This system is a method that consists of 6 semaphores (sensors), 6 stabilizers, 1 charging cable, and 1 tablet and assesses and trains the reaction time of individuals in many different environments. Before the assessments, 6 semaphores (light and sound stimuli) will be positioned to form a 180° semicircle, with each semaphore placed in increments of 45° around the semicircle.Participants will perform the test three times with 30-second intervals after one trial with their right lower-extremity, left lower-extremity, and right and left lower-extremities (random), respectively. The average of the scores obtained will be recorded and used for analysis.
Anaerobic Power | A week
  Anaerobic power test will be evaluated with the electromagnetic ergometer (Ergomedic894E, Germany). The measurement method is to adjust and set the saddle height so that the knee of each participant could have a flexion of about 5°, and thus, 0.075 kp per unit weight will be supposed to be applied when reaching one's maximum speed. Afterward, a tester in synchronization with the computer verbally count a 5-second count down following warm-up and then verbally will give a "Start" signal, after which peak anaerobic power, average power, and fatigue index will be measured while encouraging participants to perform the exercise as much as possible for 30 seconds.

CONTACTS AND LOCATIONS:
Locations (1):
- İzmir Katip Celebi University, Izmir, Turkey (Türkiye)

REFERENCES:
- [Derived] Secer E, Kaya DO. Effects of 6-Week Vibration vs. Nonvibration Foam Rolling on Performance-Related Physical Fitness Parameters in Young Male Soccer Players: A Randomized Controlled Trial. J Strength Cond Res. 2025 May 1;39(5):e647-e658. doi: 10.1519/JSC.0000000000005062. Epub 2025 Mar 4. PMID 40030119